CLINICAL TRIAL: NCT04003922
Title: Observational Study on Patients With Rasmussen Encephalitis Treated With Adalimumab: Efficacy and Tolerance in the Short and Long Term
Brief Title: Study on Patients With Rasmussen Encephalitis Treated With Adalimumab: Efficacy and Tolerance in the Short and Long Term
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-21; 2019-A00888-49 (Other: ANSM)
Record Dates: First submitted 2019-06-20; First posted 2019-07-01 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Rasmussen Encephalitis
MeSH Terms: conditions — Encephalitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Adalimumab treatment — Retrospective observational study initially and then prospective with inclusion of all the patients carrying an ER treated by Adalimumab in France. Follow-up will continue for one year if adalimumab is discontinued.

SUMMARY:
Since the initial study of cases reported between 2009 and 2015, adalimumab has become in France the immunomodulatory reference treatment used after failure of corticosteroids and immunoglobulins before a possible recourse to the hemispherotomy. This observational study is intended to document the long-term efficacy and safety of Adalimumab therapy in patients with Rasmussen encephalitis.

DETAILED DESCRIPTION:
Rasmussen Encephalitis (ER) is a particularly severe chronic inflammatory brain disorder resulting in the progressive destruction of a hemisphere. It is a rare disease although at present no precise prevalence is available. It begins preferentially in children.

This inflammatory process is accompanied by a progressive loss of function of the affected hemisphere, associated with a pharmaco-resistant partial epilepsy. The diagnosis is based on a bundle of clinical, radiological and electroencephalographic arguments. CSF analysis directs diagnosis in 50% of cases.

No anti-epileptic treatment can stop seizures. Only hemispherotomy (surgical disconnection of a cerebral hemisphere) allows it but it is associated with definitive motor and cognitive deficits.

Over the last 20 years, new therapeutic trials have focused on immuno-modulatory treatments targeted at the T-lymphocyte pathway, including tacrolimus. Although they seem to be more effective than immunoglobulins or corticosteroids, it remains transient. In addition, the number of published cases is low. In this context, starting in 2009, it has been proposed to use adalimumab (Ab anti TNF) based on:

* 1 / study of a case index
* 2 / knowledge of the pathophysiology of Rasmussen Encephalitis. To date, very few data provide precise information on the efficacy or tolerance of the use of this product in the longer term. This information is essential to confirm the place of adalimumab in the therapeutic arsenal against Rasmussen encephalitis.

Thus, in the continuation of the work carried out previously (French study on the cases between 2009 and 2015), the aim of this research projet is to complete the follow-up of the patients who previously took part in in the first study and to establish the follow-up of the patients treated by adalimumab since then.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Rasmussen Encephalitis
* Patient aged more than 2 years
* Compliant treatment with adalimumab

Exclusion Criteria:

* Patient with a differential diagnosis
* Patient suffering from Rassmussen Encephalitis but not treated with adalimumab
* Patient who has not signed the informed consent

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The implementation of a treatment with adalimumab in a patient with an ER requires the performance of a CPR within a reference center Epilepsies Rares if one complies with the rules of good clinical practice. Thus, all ER patients treated with adalimumab are referenced in a referral center. There are 7 reference centers in France, they are all partners of the study.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-04-21 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Efficiency of the treatment measured by the reduction of the number of epileptic seizures | 5 years
  The change of epileptic seizures (Will be considered as a responder patient any patient with a 50% decrease in the number of seizures between the time of inclusion and 6 months after the start of treatment). This response to treatment is re-evaluated at 12 months then every 6 months for 5 years.
Efficiency of the treatment measured by the stability if the cognitive assessment | 6 months
  Stability of the cognitive assessment: variation of less than 10 points on each of the different composite indices (QIT, ICV, IRF, IMT, IVT) of age-appropriate Weschler scales, between two cognitive assessments of 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Study Director — Assistance Publique- Hôpitaux de Marseille
Locations (16):
- France (16):
  - Chu de Bordeaux, Bordeaux
  - Chu Brest, Brest
  - Chru de Lille, Lille
  - Chu Limoges, Limoges
  - Hospices Civils de Lyon, Lyon
  - Service Neuropédiatrie, Marseille
  - Chu Montpellier, Montpellier
  - Chu de Nancy, Nancy
  - Chu Necker Ap-Hp, Paris
  - Chu Pitie Salpietriere Ap-Hp, Paris
  - Chu Robert Debre, Paris
  - Fondation Adolphe de Rothshild, Paris
  - Chu de Rennes, Rennes
  - Chu Strasbourg, Strasbourg
  - Chu Toulouse, Toulouse
  - Chru de Tours, Tours